CLINICAL TRIAL: NCT06910579
Title: Efficacy of Oxygenated Gel Therapy in the Management of Oral Aphthous Ulcers: A Randomized Controlled Clinical Trial
Brief Title: Oxygenated Gel Therapy in the Management of Oral Aphthous Ulcers
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: britishUE1
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-04

CONDITIONS: Aphthus Ulcer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): 15 patients were treated with Kenalog in orabase (Triamcinolone acetonide 0.1% oral paste 5g), four times (i.e., at 8 am, 12 noon, 4 pm, and 8 pm) a day for 7 days at intervention group.
  Interventions: Drug: topical application of Triamcinolone acetonide gel
- Oxygenated gel Group (Experimental): 15 patients who used oxygenated gel (Blue®m, Wijhe, Netherlands) were trained by the co-investigator (A.H) through real demonstration for topical application of the gel on aphthous ulcers, which entails the application of 1-2 ml of oxygenated gel directly to the ulcer two times per day and this was repeated for 7 days
  Interventions: Drug: topical application of oxygenated gel

INTERVENTIONS:
Drug: topical application of oxygenated gel — patients who used oxygenated gel (Blue®m, Wijhe, Netherlands) were trained by the co-investigator (A.H) through real demonstration for topical application of the gel on aphthous ulcers, which entails the application of 1-2 ml of oxygenated gel directly to the ulcer two times per day and this was repeated for 7 days
  Arms: Oxygenated gel Group
Drug: topical application of Triamcinolone acetonide gel — patients were treated with Kenalog in orabase (Triamcinolone acetonide 0.1% oral paste 5g), four times (i.e., at 8 am, 12 noon, 4 pm, and 8 pm) a day for 7 days at intervention group.
  Arms: control

SUMMARY:
Interventions of both groups:

Oxygenated gel Group: 15 patients who used oxygenated gel (Blue®m, Wijhe, Netherlands) were trained by the co-investigator (A.H) through real demonstration for topical application of the gel on aphthous ulcers, which entails the application of 1-2 ml of oxygenated gel directly to the ulcer two times per day and this was repeated for 7 days.

Triamcinolone acetonide Group: 15 patients were treated with Kenalog in orabase (Triamcinolone acetonide 0.1% oral paste 5g), four times (i.e., at 8 am, 12 noon, 4 pm, and 8 pm) a day for 7 days at intervention group.

Patients in both groups were reexamined after treatment at different intervals (day 3, day 5, day 7, and day 10).

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed patients with chronic aphthous stomatitis measuring ≤6 mm in size in the oral cavity and who gave written consent for participation.
* Only single ulcers were considered for the study.
* Systemically healthy patients.

Exclusion Criteria:

* The study excluded patients with a history of associated systemic disease.
* Cases of chronic aphthous stomatitis (major), lesions of herpetic form, numerous aphthae, and smoking.
* Patients with a history of hypersensitivity to the used agents.
* Pregnancy and lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 10 days
  Visual Analog Scale (0-10), which measured a range of "no pain" to "unbearable pain" on a 100 mm horizontal line [10]. to determine the intensity of pain on day 0, day 3, day 5, day 7, and day 10

SECONDARY OUTCOMES:
Size of ulcers (in mm) | 10 days
  after starting treatment, ulcer size was recorded on day 0, day 3, day 5, day 7, and day 10 using a calibrated dental probe with millimeter marking
Complete healing duration | 10 days
  the duration till complete healing is achieved is recorded in days
OHIP-14 | 10 days
  has been assessed 1 week after intervention. OHIP-14 utilizes a scale with five categories (1 = never, 2 = hardly ever, 3 = occasionally, 4 = fairly often, and 5 = very often). A lower score in any of the five categories indicates higher satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- British University in Egypt, Al Sherouk City, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared